CLINICAL TRIAL: NCT04325295
Title: Laparoscopic Ovarian Drilling Versus Gonadotrophins for Anovulatory Polycystic Ovary Syndrome Resistant to First Line Ovulation Induction: a Randomized Controlled Trial.
Brief Title: LOD vs Gn in Anovulatory PCOs Resistant to First Line Agents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Mustafa Attyia, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: induction resistant PCOs
Record Dates: First submitted 2020-03-26; First posted 2020-03-27 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Polycystic Ovary Syndrome; Anovulation
Keywords: Laparoscopic ovarian drilling; Gonadotrophins; Polycystic ovary syndrome; Anovulation; PCOs; Clomiphene resistant; Letrozole resistant
MeSH Terms: conditions — Polycystic Ovary Syndrome; Anovulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical treatment strategy: (Active Comparator)
  Interventions: Procedure: Laparoscopic ovarian drilling
- Gonadotrophins treatment strategy (Active Comparator)
  Interventions: Drug: Recombinant FSH (rFSH)

INTERVENTIONS:
Procedure: Laparoscopic ovarian drilling — LOD will be done in the follicular phase.Follow up will be done on the next cycle by performing a TVUS examination at CD 13 and measuring the dominant follicles. Ovulation is considered if a follicle reached > 17 mm and is confirmed by measuring serum progesterone at CD 21.If ovulation is not achieved in the cycle following LOD, women will be prescribed Letrozole by the dose of 2.5 mg daily for 5 days starting from CD 3, and ovulation monitoring will be done similarly. If ovulation is not achieved, the dose is increased by 2.5 mg daily in the subsequent cycle until reaching the maximum dose of 7.5 mg daily for a total of 3 cycles.With persistent resistance to Letrozole in inducing ovulation, Gn will be prescribed for 3 cycles as in Gonadotrophin strategy
  Arms: Surgical treatment strategy:
Drug: Recombinant FSH (rFSH) — A low-dose step-up protocol will be implemented. This starts on CD 3,The rFSH will be given through (IM) or(SC) injections with 75 IU and will be given once daily.Monitoring of the treatment will be done on CD 7 by TVUS and serum E2. Monitoring is individualized according to the response. Depending on the response and follicular growth, the dose may be adjusted by increasing 37.5 IU. If follicular growth failed, the dose is furtherly increased by the same amount until at least one follicle reaches 10 mm. The dose is maintained until at least one follicle reaches a diameter of 18 mm and no more than 2 follicles are bigger than 15 mm. Once reaching the desired diameter, the rFSH will be stopped and a trigger of ovulation by an IM injection of 5000 IU of hCG and sexual intercourse is encouraged on the day of trigger and the next day. Then serum P will be done 7 days after hCG injection to detect the occurrence of ovulation.
  Arms: Gonadotrophins treatment strategy

SUMMARY:
PCOS is a complex disease that is diagnosed by the presence of two of the following three: oligo/anovulation, clinical and/or biochemical hyperandrogenism, or polycystic ovaries by ultrasound . PCOS affects 4% to 21% of females in reproductive age . Although subfertility is abundant in women with PCOS, a majority of these women will achieve pregnancy naturally or by treatment.

Different treatment modalities are present for ovulation induction. Life style modifications including weight loss are encouraged for those who are overweight or obese. Pharmacological induction of ovulation represent the first line therapy for induction of ovulation. Options include aromatase inhibitors (Letrozole), Clomiphene Citrate (CC) or Metformin, alone or in combinations.

For second line treatment either Gonadotropins (Gn) or laparoscopic ovarian surgery (LOS) are the recommended options .

the objective of the trial is to study the effectiveness and safetey of surgical induction of ovulation strategy and compare it to medical induction strategy with Gonadotropins

DETAILED DESCRIPTION:
PCOS is a complex disease that is diagnosed by the presence of two of the following three: oligo/anovulation, clinical and/or biochemical hyperandrogenism, or polycystic ovaries by ultrasound . PCOS affects 4% to 21% of females in reproductive age . Although subfertility is abundant in women with PCOS, a majority of these women will achieve pregnancy naturally or by treatment.

Different treatment modalities are present for ovulation induction. Life style modifications including weight loss are encouraged for those who are overweight or obese. Pharmacological induction of ovulation represent the first line therapy for induction of ovulation. Options include aromatase inhibitors (Letrozole), Clomiphene Citrate (CC) or Metformin, alone or in combinations.

For second line treatment either Gonadotropins (Gn) or laparoscopic ovarian surgery (LOS) are the recommended options .

Systematic reviews done comparing LOD to Gn found no differences in live birth, clinical pregnancy or miscarriage rates. However, there was significant decrease in OHSS and multiple pregnancies with LOD . Giving these advantages together with being cheap, the surgical strategy may be a more favorable choice as second line treatment of anovulation . Also several randomised controlled trial (RCTs) reported normalization of ovarian reserve parameters after LOD, making it a long-lasting option compared to the one-cycle effect of medical treatment the objective of the trial is to study the effectiveness and safetey of surgical induction of ovulation strategy and compare it to medical induction strategy with Gonadotropins

ELIGIBILITY:
Inclusion Criteria:

anovulatory polycystic ovary syndrome resistant to first line ovulation induction.

* Polycystic ovary Syndrome defined by Rotterdam's criteria 2003
* Clomiphene resistance defined as failure to ovulate with a dose of 150mg per day for 5 days for 3 cycles
* Letrozole resistance defined as failure to ovulate with a dose of 7.5 mg per day for 5 days for 3 cycles

Exclusion Criteria:

* women's age < 18 years or ≥ 40 years.
* BMI > 40 kg/m2
* Patient with hyperprolactinaemia (serum prolactin above normal limits)
* Patients with hypogonadotropic hypogonadism (low serum FSH and LH)
* Patients with anovulation due to ovarian failure (serum FSH higher than normal limits)
* Male infertility
* Tubal abnormality, Known endometriosis, adenomyosis, uterine myomas or any other detected cause of female infertility
* History of ovarian surgery as laparoscopic ovarian drilling, ovarian cystectomy or oophorectomy
* History of pelvic radiation
* Patient recently treated with any type of induction of ovulation in the last three months.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Live Birth | within 12 months after of end treatment strategy
  defined as the number of births resulted in live babies after the age of viability (24th week of pregnancy)

CONTACTS AND LOCATIONS:
Overall Officials: Sayed A Abdallah, Study Director — Professor of obstetric and Gynecology,Faculty of Medicine,Assuit University O; Essam R Othman, Study Director — Assistant Professor of Obstetrics and Gynecology,Faculty of Medicine, Assuit University; Mustafa B Mohammed, Study Director — Assistant professor of Obstetrics and Gynecology, Faculty of Medicine,Assuit University; Ahmed M Alaa Eldin, Study Director — Lecturer of Obstetrics and Gynecology,Faculty of Medicine,Assuit University; Karim S Abdallah, Study Director — Assistant lecturer of Obstetrics and Gynecology,Faculty of Medicine,Assuit University

REFERENCES:
- [Background] Farquhar CM, Bhattacharya S, Repping S, Mastenbroek S, Kamath MS, Marjoribanks J, Boivin J. Female subfertility. Nat Rev Dis Primers. 2019 Jan 24;5(1):7. doi: 10.1038/s41572-018-0058-8. PMID 30679436
- [Background] Weiss NS, Kostova E, Nahuis M, Mol BWJ, van der Veen F, van Wely M. Gonadotrophins for ovulation induction in women with polycystic ovary syndrome. Cochrane Database Syst Rev. 2019 Jan 16;1(1):CD010290. doi: 10.1002/14651858.CD010290.pub3. PMID 30648738
- [Background] Lizneva D, Suturina L, Walker W, Brakta S, Gavrilova-Jordan L, Azziz R. Criteria, prevalence, and phenotypes of polycystic ovary syndrome. Fertil Steril. 2016 Jul;106(1):6-15. doi: 10.1016/j.fertnstert.2016.05.003. Epub 2016 May 24. PMID 27233760
- [Background] van Wely M, Bayram N, Bossuyt PM, van der Veen F. Laparoscopic electrocautery of the ovaries versus recombinant FSH in clomiphene citrate-resistant polycystic ovary syndrome. Impact on women's health-related quality of life. Hum Reprod. 2004 Oct;19(10):2244-50. doi: 10.1093/humrep/deh406. Epub 2004 Jul 8. PMID 15242999
- [Background] Api M. Is ovarian reserve diminished after laparoscopic ovarian drilling? Gynecol Endocrinol. 2009 Mar;25(3):159-65. doi: 10.1080/09513590802585605. PMID 19347705
- [Background] Debras E, Fernandez H, Neveu ME, Deffieux X, Capmas P. Ovarian drilling in polycystic ovary syndrome: Long term pregnancy rate. Eur J Obstet Gynecol Reprod Biol X. 2019 Aug 13;4:100093. doi: 10.1016/j.eurox.2019.100093. eCollection 2019 Oct. PMID 31497757
- [Background] Amer SA, Banu Z, Li TC, Cooke ID. Long-term follow-up of patients with polycystic ovary syndrome after laparoscopic ovarian drilling: endocrine and ultrasonographic outcomes. Hum Reprod. 2002 Nov;17(11):2851-7. doi: 10.1093/humrep/17.11.2851. PMID 12407038
- [Background] Farquhar C, Brown J, Marjoribanks J. Laparoscopic drilling by diathermy or laser for ovulation induction in anovulatory polycystic ovary syndrome. Cochrane Database Syst Rev. 2012 Jun 13;(6):CD001122. doi: 10.1002/14651858.CD001122.pub4. PMID 22696324
- [Background] Nahuis MJ, Oude Lohuis E, Kose N, Bayram N, Hompes P, Oosterhuis GJ, Kaaijk EM, Cohlen BJ, Bossuyt PP, van der Veen F, Mol BW, van Wely M. Long-term follow-up of laparoscopic electrocautery of the ovaries versus ovulation induction with recombinant FSH in clomiphene citrate-resistant women with polycystic ovary syndrome: an economic evaluation. Hum Reprod. 2012 Dec;27(12):3577-82. doi: 10.1093/humrep/des336. Epub 2012 Sep 20. PMID 23001778